CLINICAL TRIAL: NCT01101360
Title: Evaluation of Fractional Radiofrequency (Matrix RF) Stand Alone and Combined With PDL Treatment on Port Wine Stains
Brief Title: Port Wine Stains Treatment Matrix RF Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DC75761
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Port Wine Stains
Keywords: port wine stains; radiofrequency; Pulse Dye Laser
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Matrix RF followed by Pulse Dye Laser (Active Comparator)
  Interventions: Device: Matrix RF; Device: Matrix RF followed by Pulse Dye Laser; Device: Pulse Dye Laser followed by Matrix RF

INTERVENTIONS:
Device: Matrix RF — Section of port wine stain to be treated 5 times every 5 weeks (+/- 1 week)
Device: Matrix RF followed by Pulse Dye Laser — Section of port wine stain to be treated 5 times every 5 weeks (+/- 1 week)
Device: Pulse Dye Laser followed by Matrix RF — Section of port wine stain to be treated 5 times every 5 weeks (+/- 1 week)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the Matrix RF for Port Wine Stains based on clinical and histological analyses.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy males or females older than 18 to 65 years of age.
* Having a low to mid depth Port Wine Stain of at least 5 cm2.
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* PWS on lower legs or hands.
* Pregnant and/or breastfeeding.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* Having a permanent implant in the treated area, such as an injected chemical substance in the face (if treated).
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
* Use of retinoids, antioxidants or medical grade of skin nourishing supplements within 2 months of treatment or during the study.
* Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study (if face is treated).
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received Botox/collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months of treatment or during the study (if face is treated).
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study (if face is treated).
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: active acne, excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including actinic keratosis, presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* Tattoo or permanent make-up in the treated area.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within three month prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Time to complete healing | Up to 30 weeks
  Assess safety of the Matrix RF treatment for port wine stains
Adverse events recording and monitoring | Up to 40 weeks

SECONDARY OUTCOMES:
Clearance of port wine stain | Up to 40 weeks
Lightening of the port wine stain | Up to 40 weeks
  Evaluation of lightening of the port wine stain will be made with reflectance spectrophotometer at all treatments and at 6 and 12 weeks following the last treatment.
Improvement of port wine stain | Up to 30 weeks
  Assessment to be done by the subject via subject questionnaire during these visits
Reduction in blood vessel concentration | Up to 40 weeks
  Biopsies taken from consenting subjects at one of the time points will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States